CLINICAL TRIAL: NCT05590429
Title: Frequency and Complications of Blood Transfusion in Patients With Lung Cancer
Brief Title: Blood Transfusion in Patients With Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Olcay Ayçiçek, Assistant professor, Karadeniz Technical University
Other Study IDs: 24237859-782
Record Dates: First submitted 2021-06-13; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-04

CONDITIONS: Transfusion-Transmitted Infection
Keywords: Hemoglobin, lung canser, complication
MeSH Terms: conditions — Transfusion Reaction | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood transfusion — No intervention

SUMMARY:
The main purpose of approaching the anemic patient is to provide and maintain hemoglobin levels that will allow oxygen to reach the tissue at an adequate level. This critical level may vary from patient to patient, the age of the patient and other accompanying diseases are among the determining factors. The most important factor in transfusion indication is the insufficiency of cardiopulmonary compensation mechanisms due to anemia in the patient and the patient becoming symptomatic. Red blood cell (RBC) transfusions are common in the treatment of cancer patients.

In cancer patients, similar to other patient populations, the indication for RBC transfusion is to alleviate anemia, which is actually symptomatic. However, the decision to transfuse should not be guided solely by the hemoglobin concentration.

With this study, it is aimed to develop clinical practices to prevent unnecessary transfusion practices in lung cancer patients, to encourage the application of other supportive treatment options, and to take preventive measures before anemia develops

DETAILED DESCRIPTION:
Blood is a living tissue composed of specific structures, each with distinct functions. Blood transfusion is a tissue or even organ transplantation. Unnecessary blood transfusion should not be done, and the missing component should be replaced in the patient.

The need for transfusion seen in medical diseases is often in the form of chronic anemia, except for a few conditions that cause sudden bleeding. Repeated transfusions may be required in these patients during the course of their disease and related problems may arise. For this reason, while determining the indication for transfusion, it is absolutely necessary to perform the benefit-harm analysis correctly.

The main purpose of approaching the anemic patient is to provide and maintain hemoglobin levels that will allow oxygen to reach the tissue at an adequate level. This critical level may vary from patient to patient, the age of the patient and other accompanying diseases are among the determining factors. The most important factor in transfusion indication is the insufficiency of cardiopulmonary compensation mechanisms due to anemia in the patient and the patient becoming symptomatic. Red blood cell (RBC) transfusions are common in the treatment of cancer patients.

Generally, patients with oncological and hematological malignancies use approximately 34% of the RBC source. In cancer patients, similar to other patient populations, the indication for RBC transfusion is to alleviate anemia, which is actually symptomatic. However, the decision to transfuse should not be guided solely by the hemoglobin concentration. No single criterion can be used as an indicator of RBC transfusion.

The clinical condition of the patient must be taken into account. Anemia can be seen in approximately 90% of patients during chemotherapy treatment. Cytotoxic drugs often cause the loss, destruction and reduction of RBCs that cause anemia. Especially lung and gynecological cancers are highly associated with anemia. Platinum-based chemotherapeutics are often preferred in the treatment of such cancers. Anemia in cancer can reduce quality of life and increase cancer-related fatigue and may be a poor indicator of clinical outcomes. That is why, in clinical practice, transfusions are often performed in cancer patients.

In general, a hemoglobin level of 7 g / dL is a suitable indicator for red blood cell (RBC) transfusion in stable patients without complications. However, patients with cardiovascular disease or acute coronary syndrome can be transfused at a hemoglobin level of 8 g / dL.

Although the indications for transfusion in patients with other types of complications are unclear, cancer patients have reported improved clinical well-being when kept at about 7 g / dL in hemoglobin levels, but no study results suggested an absolute hemoglobin level that is optimal for patients with cancer.

With this study, it is aimed to develop clinical practices to prevent unnecessary transfusion practices in lung cancer patients, to encourage the application of other supportive treatment options, and to take preventive measures before anemia develops.

Patients who have been followed up and receiving chemotherapy in our chest diseases department in the last 5 years will be included in our study. Patients who were diagnosed with lung cancer between 01/01 / 2014-31 / 12/2018, followed up in the chest diseases service and given chemotherapy will be included in the study. Patient data will be retrospectively collected using file records and hospital automation system (clinical course, blood bank data, consultation records, etc.). The study will begin after the approval of the ethics committee and will continue for 6 months.

Exclusion Criteria; Patients with known hematological malignancies other than lung cancer, patients who were diagnosed with anemia before chemotherapy treatment, who received treatment for this reason, patients who were diagnosed with lung cancer in our clinic but did not continue chemotherapy treatment in our clinic afterwards, and patients who are thought to impair data integrity due to incomplete data will be excluded from the study.

Patients' data to be followed; Exclusion Criteria; Patients with known hematological malignancies other than lung cancer, patients who were diagnosed with anemia before chemotherapy treatment, who received treatment for this reason, patients who were diagnosed with lung cancer in our clinic but did not continue chemotherapy treatment in our clinic afterwards, and patients who are thought to impair data integrity due to incomplete data will be excluded from the study.

Patients' data to be followed; Demographic characteristics, comorbid diseases, cancer type and stage, how long it was followed up with this diagnosis, Hb value before starting chemotherapy, whether RBC transfusion was performed during the follow-up period, which Hb value of blood transfusion was applied, how many units of RBC or other blood were taken during the follow-up period. product replacement, how many cures of chemotherapy they received in total, which chemotherapy drugs they took, whether there was a delay in treatment due to treatment-related anemia, the most frequent indications and complications of transfusion (allergic reaction, febrilereax., infection and thromboembolic complications), whether they received additional radiotherapy. , whether they received GMC-SF due to anemia, blood groups, survival times, how many times there was cancer progression under treatment, and if there is distant metastasis, the location of metastasis was aimed to be screened.

In the analysis of the data; The compliance of the data to normal distribution will be examined by Shapiro Wilk and Kolmogorog Smirnov tests. Kruskall-Wallis, Mann-Whitney U, student-t and chi-square tests will be used for comparisons between groups. General linner modeling, Wilcowon and Friedman tests will be used in serially tracked data. Data will be given as percentage, mean (std deviation) and median (minimum-maximum). The chi-square test will be used to compare qualitative data. Categorical data will be presented in the form of frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age diagnosed with non-small cell lung cancer Patients over 18 years of age diagnosed with small cell lung cancer Patients diagnosed with lung cancer and undergoing chemotherapy

Exclusion Criteria:

Patients with known hematological malignancies other than lung cancer, patients who were diagnosed with anemia before chemotherapy treatment, who received treatment for this reason, patients who were diagnosed with lung cancer in our clinic but did not continue chemotherapy treatment in our clinic afterwards, patients who are thought to impair data integrity due to missing data will be excluded from the study

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with lung cancer and treated
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-11-02 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
evaluate the relationship between blood transfusion frequency and disease prognosis | 01.10.2020-01.06.2022
  With this study, it is aimed to develop clinical practices to prevent unnecessary transfusion practices in lung cancer patients, to encourage the application of other supportive treatment options and to take preventive measures before anemia develops.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Küçük, MD, Study Chair — Department of Chest Diseases, Division Of Intensive Care Medicine, Faculty of Medicine, Karadeniz Technical University; A. Oguzhan Küçük, MD, Study Chair — Department of Chest Diseases, Division Of Intensive Care Medicine, Faculty of Medicine, Karadeniz Technical University; Merve Algın, MD, Study Chair — Department of Chest Diseases, Faculty of Medicine, Karadeniz Technical University; Ayşegul Pehlivanlar, MD, Study Chair — Department of Chest Diseases, Faculty of Medicine, Karadeniz Technical University; Funda Öztuna, Prof, Study Chair — Department of Chest Diseases, Faculty of Medicine, Karadeniz Technical University; Olcay Ayçiçek, Principal Investigator — Department of Chest Diseases, Faculty of Medicine, Karadeniz Technical University
Locations (1):
- Department of Chest Diseases, Division Of Intensive Care Medicine, Faculty of Medicine, Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No